CLINICAL TRIAL: NCT03248193
Title: Concomitant Limb Cryocompression and Scalp Cooling to Reduce Paclitaxel-induced Neuropathy and Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2017/00138
Record Dates: First submitted 2017-08-01; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)
Keywords: paclitaxel; neuropathy; hypothermia; cryocompression; alopecia
MeSH Terms: conditions — Hypothermia; Alopecia

STUDY DESIGN:
Intervention Model Description: This study will consist of two parts:
  A) Healthy subjects: To assess safety and tolerability of scalp and limb hypothermia, as well as to determine the optimal temperature and pressure to be used. Establishing the occurrence or lack of core hypothermia will be studied.
  B) Cancer patients: Once the optimal temperature and pressure of scalp and limb hypothermia is established in healthy patients, a group of cancer patients will undergo concomitant scalp and limb hypothermia over multiple cycles of chemotherapy to establish safety and tolerability of repeated therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental): To assess safety and tolerability of scalp and limb hypothermia, as well as to determine the optimal temperature and pressure to be used. Establishing the occurrence or lack of core hypothermia will be studied.
  Interventions: Device: Concomitant limb cryocompression and scalp cooling
- Cancer subjects (Experimental): Once the optimal temperature and pressure of scalp and limb hypothermia is established in healthy patients, a group of cancer patients will undergo concomitant scalp and limb hypothermia over multiple cycles of chemotherapy to establish safety and tolerability of repeated therapy.
  Interventions: Device: Concomitant limb cryocompression and scalp cooling

INTERVENTIONS:
Device: Concomitant limb cryocompression and scalp cooling — Part 1: Establishing optimal temperature for hypothermia therapy. Healthy subjects will undergo 3 hours of cryocompression various temperature levels.
  Part 2: Establishing optimal pressure for hypothermia therapy. Each subject will undergo cryocompression (fixed at the lowest tolerated temperature established in Section 1) over 3 hours. The pressure ranges to be tested are either low, medium, or high.
  Part 3: Establishing safety and tolerability of scalp hypothermia. Scalp hypothermia will be administered over 3 hours using the cooling cap attached to the cooling device.
  Part 4: Establishing safety and tolerability of concomitant therapy. Subjects will undergo simultaneous scalp hypothermia and four-limb cryocompression at the temperature and pressure established in Sections 1 and 2. The concomitant therapy will be administered over 3 hours.
  Arms: Healthy subjects
Device: Concomitant limb cryocompression and scalp cooling — The study population will comprise of cancer patients scheduled to receive weekly paclitaxel chemotherapy for a maximum of 12 cycles.
  Paclitaxel will be administered as a one-hour infusion. Concomitant scalp cooling and limb cryocompression sessions comprised of a pre-cooling period (one hour), continued with paclitaxel infusion and a post-cooling period (on average 30 minutes after the end of paclitaxel infusion). Overall, hypothermia will be administered for no longer than four hours.
  Cryocompression will be administered on patients based on the lowest tolerated temperature and optimal pressure as determined in healthy subjects.
  Arms: Cancer subjects

SUMMARY:
Paclitaxel is a chemotherapy drug that is used to treat breast cancer, one of the most common cancers. It causes two side effects very often - hair-loss and numbness. Until recently, there have been no known ways to prevent or treat either side effect. Recently, cooling of the scalp to prevent hair loss caused by paclitaxel was approved. Our team is developing a method to prevent numbness caused by paclitaxel by using a device that cools the arms and the legs, while applying mild pressure, and this technique is called cryocompression. As scalp cooling use in day-to-day cancer care increases, future studies involving cryocompression to treat neuropathy must take this into account, lest patients be denied or are required to trade-off one treatment for the other. However, there is concern of causing a reduction in core body temperature, which would not be safe or a general intolerance to this treatment. Both scalp cooling and limb cryocompression individually have not shown to cause this, but simultaneous use has not been studied previously. Clinical safety studies, in healthy subjects and cancer patients would need to be conducted to prove this theory, which is being proposed by currently.

DETAILED DESCRIPTION:
Paclitaxel is a key chemotherapeutic agent used in the management of common cancers, such as breast cancer. Chemotherapy-induced peripheral neuropathy (CIPN) due to paclitaxel is a common dose-limiting toxicity with no effective prevention or treatment. Limb cryocompression is currently being developed as a method to reduce CIPN. Another common toxicity of paclitaxel is chemotherapy induced alopecia (CIA), for which scalp-cooling is currently an approved therapy to reduce the incidence of this adverse effect. As scalp cooling use in day-to-day clinical practice increases, future studies involving hypothermia to treat neuropathy must factor this into the treatment algorithm, lest patients be denied or are required to trade-off one treatment for the other. However, there is concern of causing core hypothermia and/or general intolerance to concomitant therapy. Both scalp-cooling and cryocompression individually have not shown to cause this, but simultaneous use has not been studied previously. Clinical safety studies, in healthy subjects and cancer patients would need to be conducted first, before larger efficacy studies are performed. We propose that we can deliver scalp-cooling and limb cryocompression with a single treatment modality to prevent two toxicities of paclitaxel - CIA and CIPN. This study will consist of two parts: A) Healthy subjects: To assess safety and tolerability of scalp and limb cryocompression, as well as to determine the optimal temperature and pressure to be used, that will contribute to the cryocompression protocol. The occurrence of core hypothermia or intolerance will be closely monitored B) Cancer patients: Once the optimal cryocompression protocol is established in healthy patients, a group of cancer patients will undergo concomitant limb cryocompression and scalp cooling over multiple cycles of chemotherapy to establish safety and tolerability of repeated therapy. Early clinical efficacy signal data will also be collected, to prepare for the subsequent larger randomized efficacy study.

ELIGIBILITY:
The inclusion criterion for the healthy subjects:

* Age 21-80 years
* Signed informed consent from patient.
* No history of neuropathy
* ECOG 0
* No history of hospitalization in the past 6 months

The inclusion criteria for the cancer patients:

* Age 21- 80 years.
* Signed informed consent from patient
* Scheduled to receive weekly paclitaxel chemotherapy

For both healthy subjects and cancer patients:

* Open skin wound or ulcers of the limbs
* A score of more than 5 in the Total Neuropathy Score (TNS) at baseline (see outcome parameters) (Not applicable for healthy subjects)
* History of Raynaud's phenomenon, peripheral vascular disease, or poorly controlled diabetes

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Investigation of safety and tolerability of concomitant scalp cooling and limb cryocompression in healthy subjects: defined as the number of patients with treatment-related intolerance as assessed by CTCAE v4.0 and tolerability scales | From the start of assessment until study completion, an average of 1 year
Investigation of safety and tolerability of concomitant scalp cooling and limb cryocompression in cancer patients: defined as the number of patients with treatment-related intolerance as assessed by CTCAE v4.0 and tolerability scales. | From the start of assessment until study completion, an average of 1 year

SECONDARY OUTCOMES:
Difference in sensory nerve action potential on nerve conduction tests before and at the end of taxane-based chemotherapy with limb cryocompression. | From the start of assessment until study completion, an average of 2 years
Difference in qualitative symptom scores before and at the end of taxane-based chemotherapy with limb cryocompression. | From the start of assessment until study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Raghav Sundar, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Windebank AJ, Grisold W. Chemotherapy-induced neuropathy. J Peripher Nerv Syst. 2008 Mar;13(1):27-46. doi: 10.1111/j.1529-8027.2008.00156.x. PMID 18346229
- [Background] Sundar R, Bandla A, Tan SS, Liao LD, Kumarakulasinghe NB, Jeyasekharan AD, Ow SG, Ho J, Tan DS, Lim JS, Vijayan J, Therimadasamy AK, Hairom Z, Ang E, Ang S, Thakor NV, Lee SC, Wilder-Smith EP. Limb Hypothermia for Preventing Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients: A Pilot Study. Front Oncol. 2017 Jan 10;6:274. doi: 10.3389/fonc.2016.00274. eCollection 2016. PMID 28119855
- [Background] Bandla A, Sundar R, Liao LD, Sze Hui Tan S, Lee SC, Thakor NV, Wilder-Smith EP. Hypothermia for preventing chemotherapy-induced neuropathy - a pilot study on safety and tolerability in healthy controls. Acta Oncol. 2016;55(4):430-6. doi: 10.3109/0284186X.2015.1075664. Epub 2015 Sep 11. PMID 26360921